CLINICAL TRIAL: NCT00210535
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Topiramate for the Prophylaxis of Migraine in Pediatric Subjects 12 to 17 Years of Age
Brief Title: A Study of the Effectiveness and Safety of Topiramate for the Prevention of Migraine Attacks in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR002245
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-01

CONDITIONS: Migraine; Vascular Headaches
Keywords: Topiramate; Migraine; Migraine headache; Migraine prevention; Pediatric
MeSH Terms: conditions — Migraine Disorders; Vascular Headaches | interventions — Topiramate

INTERVENTIONS:
Drug: Topiramate; Placebo

SUMMARY:
The primary purpose of this study is to evaluate the effectiveness and safety of topiramate compared with placebo in the prevention of migraine attacks in children (12 to 17 years of age).

DETAILED DESCRIPTION:
This is an outpatient, randomized, double-blind, placebo-controlled study to evaluate the effectiveness of 2 dosages of topiramate (50 and 100 milligrams/day) compared with placebo in the prevention of migraine attacks in children 12 to 17 years of age. The study is composed of 3 phases: pretreatment, double-blind treatment for 4 months (16 weeks), and posttreatment. During the study, patients will maintain headache and medication records to document the following: occurrence and duration of headaches; severity of headache pain; whether or not the headache is pulsating or aggravated by physical activity; associated symptoms, such as nausea, vomiting, photophobia, phonophobia, abdominal pain; and medication taken to relieve headache pain or symptoms. Assessment of efficacy include the percent reduction in the frequency of monthly migraine attacks over the last 12 weeks of the double-blind treatment phase compared with prospective BL period. In addition, the percent reduction in (a) average monthly migraine days, (b) average monthly headache days, and (c) monthly migraine rate, over the last 12 weeks of the double-blind treatment phase compared with the pretreatment phase will be assessed. Safety assessments include the incidence of adverse events, measurement of vital signs (pulse, blood pressure, oral temperature), results of pregnancy tests, physical and neurologic examinations, clinical laboratory tests (hematology, biochemistry, and urinalysis), and monitoring for visual or ocular disturbances, heat intolerance, renal or urinary disturbance, depression and rash. The study hypothesis is that the percent reduction in frequency of monthly (28-day) migraine attacks (using the 48-hour rule) from the prospective baseline period (pretreatment phase) to the last 12 weeks of the double-blind phase will be significantly better for the topiramate groups than for the placebo group. Topiramate tablets (25 milligrams) or placebo, beginning at 25mg once daily (Week 1), increasing to twice daily total of 50mg or 100mg (Week 4). Maximum dosage of topiramate (or placebo) continues for next 12 weeks. Dosage may be reduced once at investigator's discretion.

ELIGIBILITY:
Inclusion Criteria:

* History of migraine (with or without aura) conforming to International Headache Society (IHS) criteria for pediatric subjects for >=6 months prior to screening
* Requires migraine prophylactic therapy, and if previously treated to prevent attacks, had unsatisfactory response to therapy
* Experienced an average of 3 to 12 migraine attacks and no more than 14 headache days per month during the 3 months prior to the study
* Females must be sexually abstinent, surgically sterile, or using adequate contraceptive measures, and have negative pregnancy tests before and during the study

Exclusion Criteria:

* Currently taking or previously unable to tolerate topiramate, or previously failed therapy with topiramate for migraine prophylaxis
* Has mixed headaches and is unable to distinguish migraines from other headache types
* Overuses pain medications or specific agents for abortive treatment of migraine attacks
* Has a body mass index (BMI) greater than 40 or weighs more than 200 pounds, or is markedly underweight (below 5th percentile) for his or her age

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2005-06; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Percent reduction in the frequency of monthly migraine attacks (using 48-hour rule) over the last 12 weeks of the double-blind treatment phase compared with the 4-week prospective baseline period.

SECONDARY OUTCOMES:
Percent reduction in (a) average monthly migraine days, (b) average monthly headache days, and (c) monthly migraine rate, over the last 12 weeks of the double-blind treatment phase compared with the prospective baseline period.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Topiramate for the Prophylaxis of Migraine in Pediatric Subjects 12 to 17 Years of Age — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=463&filename=CR002245_CSR.pdf